CLINICAL TRIAL: NCT01115309
Title: XprESS Registry Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1677-001
Record Dates: First submitted 2010-04-29; First posted 2010-05-04 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Sinusitis
Keywords: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- XprESS Balloon Device (Other): Sinus dilation
  Interventions: Device: XprESS Balloon Device

INTERVENTIONS:
Device: XprESS Balloon Device — Sinus dilation completed with the XprESS Balloon Device with or without additional endoscopic sinus surgery procedures (dilation of the frontal recesses, maxillary ostia, and/or sphenoid sinus ostia).

SUMMARY:
This is a prospective, non-randomized, multi-center study to assess safety and long-term patency of the ostia treated with the XprESS device per the device indication for use (IFU).

DETAILED DESCRIPTION:
Endoscopic balloon-only and hybrid-balloon procedures involving dilation of the frontal recesses, maxillary ostia, and/or sphenoid sinus ostia were performed in 175 patients.

One-month follow-up was required for all patients. The first 50 patients enrolled also consented to a 1-year follow-up. Complications and sinus symptom severity were assessed at the 1-month visit. Symptom severity and ostial patency of the treated sinuses were evaluated at the 1-year visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Scheduled to undergo sinus surgery with planned use of the XprESS Balloon Device consistent with the tool's Indication for Use
* Willing and able to provide consent

Exclusion Criteria:

* Known Samter's Triad
* History of primary ciliary dysfunction
* History of cystic fibrosis
* Known to be immunosuppressed
* Hemophilia
* Currently enrolled in another pre-approval investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Grebner, Study Chair — Entellus Medical
Locations (1):
- Texas Sinus Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brodner D, Nachlas N, Mock P, Truitt T, Armstrong M, Pasha R, Jung C, Atkins J. Safety and outcomes following hybrid balloon and balloon-only procedures using a multifunction, multisinus balloon dilation tool. Int Forum Allergy Rhinol. 2013 Aug;3(8):652-8. doi: 10.1002/alr.21156. Epub 2013 Feb 19. PMID 23424023

RESULTS

PARTICIPANT FLOW:
Period: Procedure Safety (1-Month)
Arm/Group | XprESS Balloon Device
Started | 175
Completed | 172
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Period: Long-term Follow-up
Arm/Group | XprESS Balloon Device
Started | 50
6-Month Follow-up | 46
12-Month Follow-up | 44
Completed | 44
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | XprESS Balloon Device
Number analyzed (Participants) | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 97
Region of Enrollment [Number; unit: participants]
  United States | 175
Lund-Mackay score [Mean (Standard Deviation); unit: units on a scale] — The Lund-Mackay score is a method to grade CT scan findings of the paranasal sinuses and ostiomeatal complex for chronic rhinosinusitis. Each sinus and ostiomeatal complex on each side is scored as 0 (no abnormality), 1 (partial opacification) or 2 (complete opacification). The ostiomeatal complex is assigned a score of either 0 (not obstructed) or 2 (obstructed). An aplastic frontal sinus is assigned a score of 0. The Lund-Mackay score can range from 0 to 24 with higher values indicating greater disease severity. Population: Lund-Mackay is provided for those participants who had a preoperative scan available.
  units on a scale
    number analyzed (Participants) | 86
    (all) | 6.9 (4.6)
SNOT-20 [Mean (Standard Deviation); unit: units on a scale] — The 20-item Sino-Nasal Outcome Test (SNOT-20) is a validated, patient-reported outcome assessment to measure the presence and severity of symptoms of chronic rhinosinusitis. Each symptom is scored from 0 (no problem) to 5 (as bad as it can be). The overall score is the mean of the 20 individual items, with a range from 0 to 5 with higher scores indicating greater disease severity. A difference of 0.8 has been determined to be the minimal clinically important difference (MCID) for the SNOT-20. Population: Baseline SNOT-20 assessments were inadvertently lost for 5 participants.
  units on a scale
    number analyzed (Participants) | 170
    (all) | 2.1 (1.0)
Nasal polyps [Count of Participants; unit: Participants] — Number of participants with nasal polyps.
  Participants | 55
Area of sinusitis [Count of Participants; unit: Participants] — Number of participants with disease in the applicable sinus.
  Participants
    Maxillary | 162
    Anterior ethmoid | 133
    Posterior ethmoid | 116
    Frontal | 145
    Sphenoid | 106

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessments
Description: Adverse event reporting as related to XprESS device or procedure
Time Frame: 1 month after procedure
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | XprESS Balloon Device
Number analyzed (Participants) | 175
Participants | 2

2. Secondary Outcome: Sino-Nasal Outcome Test (SNOT-20) at 1 Month
Description: The 20-item Sino-Nasal Outcome Test (SNOT-20) is a validated, patient-reported outcome assessment to measure the presence and severity of symptoms of chronic rhinosinusitis. Each symptom is scored from 0 (no problem) to 5 (as bad as it can be). The overall score is the mean of the 20 individual items, with a range from 0 to 5 with higher scores indicating greater disease severity. A difference of 0.8 has been determined to be the minimal clinically important difference (MCID) for the SNOT-20.
Time Frame: Baseline and 1 month after procedure
Population: All participants with baseline and 1-month SNOT-20 scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | XprESS Balloon Device
Number analyzed (Participants) | 170
score on a scale
  Baseline | 2.1 (1.0)
  1-Month Follow-up | 1.0 (0.8)
Statistical Analysis 1: Comparison: XprESS Balloon Device; Test type: Superiority; p < 0.0001, t-test, 2 sided — Paired t-tests were used to evaluate whether the change in outcomes from baseline to follow-up were statistically different from zero. A p value <0.05 is considered statistically significant

3. Secondary Outcome: SNOT-20 at 6 Months
Description: as for outcome 2
Time Frame: Baseline and 6 months post procedure
Population: Participants enrolled in the long-term follow-up who have matching baseline and 6-month SNOT-20 scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- XprESS Balloon Device Long-term Follow-up: Fifty participants who were enrolled in the long-term follow-up.
Arm/Group | XprESS Balloon Device Long-term Follow-up
Number analyzed (Participants) | 46
score on a scale
  Baseline | 2.0 (1.1)
  6-Month Follow-up | 0.8 (0.7)
Statistical Analysis 1: Comparison: XprESS Balloon Device Long-term Follow-up; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: SNOT-20 at 12 Months
Description: as for outcome 2
Time Frame: Baseline and 12 months post procedure
Population: Participants who were enrolled in the long-term follow-up and have matching baseline and 12-month SNOT-20 scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | XprESS Balloon Device Long-term Follow-up
Number analyzed (Participants) | 44
score on a scale
  Baseline | 1.9 (1.1)
  12-Month Follow-up | 0.8 (0.7)

5. Other Pre Specified Outcome: Number of Sinuses Demonstrating Functional Patency
Description: Functional patency of the sinus ostia originally treated with XprESS was assessed by the clinical site either by visual endoscopic evidence of a clear drainage path or radiographic evidence of a completely aerated sinus at 12-month follow-up for the first 50 patients treated in the study.
Time Frame: 12 months post procedure
Population: Frontal and sphenoid sinuses treated with XprESS and evaluated by endoscopy or CT scan at 12 months post procedure.
Measure: Count of Units; unit: Sinuses
Units Other Than Participants: Sinuses
Arm/Group | XprESS Balloon Device Long-term Follow-up
Number analyzed (Participants) | 44
Number analyzed (Sinuses) | 83
Sinuses | 76

ADVERSE EVENTS:
Time Frame: Adverse events from time of procedure through 12 months post procedure. Per protocol, only 50 of the 175 enrolled participants were followed after the 1-month postprocedure visit.
Arm/Group | XprESS Balloon Device
All-Cause Mortality (participants affected / at risk) | 0/175
Serious Adverse Events (participants affected / at risk) | 0/175
Other Adverse Events (participants affected / at risk) | 0/175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less